CLINICAL TRIAL: NCT06045403
Title: Early-warning Intervention for Heat and Cold in Older Hypertensive Patients: Impact on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tiantian Li (Other Government)
Responsible Party: Sponsor-Investigator, Tiantian Li, professor, Centers for Disease Control and Prevention, China
Organization: Centers for Disease Control and Prevention, China (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202381
Record Dates: First submitted 2023-09-10; First posted 2023-09-21 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Cold Temperature; epicatechin gallate; Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combined intervention (Experimental): Participants in the combined intervention group will receive real-time health risk warnings for heat waves and cold spells via a WeChat mini-program and will perform daily self-monitoring of BP and ECG using automated home devices.
  Interventions: Behavioral: Issuing health risk warning for a heat or cold; Device: A digital heat or cold health risk early warning tool; Behavioral: Perform daily self-monitoring of their BP and ECG; Device: Self-monitoring blood pressure and ECG device
- Self-monitoring alone (Experimental)
  Interventions: Behavioral: Perform daily self-monitoring of their BP and ECG; Device: Self-monitoring blood pressure and ECG device
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Issuing health risk warning for a heat or cold — Whenever a health risk warning for a heat or cold is issued, only the elderly in the combined intervention group will be alerted to the early warning information through the digital heat or cold health risk early warning tool.
  Arms: Combined intervention
Device: A digital heat or cold health risk early warning tool — A WeChat mini-program provides real-time updates on early warnings and health advisories.
  Arms: Combined intervention
Behavioral: Perform daily self-monitoring of their BP and ECG — Participants in the self-monitoring alone group were instructed to self-measure their BP three times each morning (from 6:00 a.m. to 8:00 a.m.) and evening (from 6:00 p.m. to 8:00 p.m.) at home, and to self-administer ECG measurements twice during the same morning and evening timeframes.
  Arms: Combined intervention; Self-monitoring alone
Device: Self-monitoring blood pressure and ECG device — Devices for self-monitoring blood pressure and electrocardiography (ECG).
  Arms: Combined intervention; Self-monitoring alone

SUMMARY:
This cluster-randomized trial, conducted in Tianjin, China, aims to evaluate the effectiveness of integrating a digital health risk early warning tool for heat with self-monitoring. Additionally, the study assesses the effectiveness of combining a digital health risk early warning tool for cold with self-monitoring. Communities from three districts will be randomly assigned to one of three groups: the combined intervention group, the self-monitoring group, and the control group. The primary objective of the study is to evaluate the effectiveness of the intervention in improving sleep quality, as well as understanding its underlying biological mechanisms.

DETAILED DESCRIPTION:
This cluster-randomized trial will be conducted in various districts across Tianjin, China. As part of the early warning interventions for heat waves and cold spells, three communities from each of the two selected districts will be randomly chosen and assigned to one of three groups: the combined intervention group, the self-monitoring group, or the control group. The study will be divided into pre-intervention and intervention phases. The pre-intervention period for the heat wave health early-warning information intervention spans from July 1st, 2023, to July 7th, 2023, followed by the intervention period from July 8th to September 9th, 2023. Similarly, during the cold spell health early-warning information intervention, the pre-intervention phase occurs from December 1st, 2023, to December 7th, 2023, and the intervention.

Participants in the combined intervention group will receive heat health risk warnings via digital tools, specifically a WeChat mini-program, providing real-time updates on early warnings and health advisories. Additionally, they will be instructed to perform daily self-monitoring of their blood pressure (BP) and electrocardiogram (ECG) using automated home devices. Participants in the self-monitoring alone group will engage in daily BP and ECG monitoring but not receive any health warnings. In contrast, the control group will monitor their BP and ECG only during baseline assessments and routine health check-ups (the day after the first heat wave in July and August 2023, as well as following the first cold spell in January and February 2024).

All participants will be required to record their daily time-activity patterns. During the baseline and subsequent check-ups, data will be collected on participants' demographics, medical history, lifestyle factors (e.g., diet, smoking, physical activity), environmental exposures, sleep quality, mental health status (including stress levels, emotional stability, and psychological resilience), medication adherence, cardiovascular and cerebrovascular symptoms, respiratory system symptoms, and perceptions of heatwaves and cold spells. In addition, blood, urine, and stool samples will be gathered for further analysis.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 60 to 65 years Individuals with a diagnosis of hypertension Individuals with untreated blood pressure above 140/90 mm Hg

Exclusion Criteria:

Having a history of coronary heart disease, heart failure, or stroke Unable to cooperate with follow-up

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the PSQI score | baseline, six months
  The PSQI score is measured by the pittsburgh sleep quality index questionnaire. The PSQI consists of 19 individual items that assess seven key components of sleep: subjective sleep quality, sleep latency (the time it takes to fall asleep), sleep duration, habitual sleep efficiency (the ratio of total sleep time to time spent in bed), sleep disturbances, use of sleep medication, and daytime dysfunction.Each of the seven components is scored from 0 to 3, with the total PSQI score ranging from 0 to 21. A total score greater than 5 indicates poor sleep quality, while a lower score suggests good sleep quality.

SECONDARY OUTCOMES:
Change from baseline in the control rate of blood pressure (SBP/DBP <140/90 mm Hg) | baseline, six months
  The blood pressure was measured by a self-monitored electronic sphygmomanometer (Model Maibobo, Shenzhen Yike Network Technology Co., Ltd., China). The proportion of participants achieving a systolic blood pressure (SBP) below 140 mm Hg and a diastolic blood pressure (DBP) below 90 mm Hg is calculated by dividing the number of participants who meet these criteria by the total number of participants at baseline and each routine health check-up.
Change from baseline in the risk of the overall warning level for abnormal ECG. | baseline, six months
  Overall warning level for abnormal ECG is measured by a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China). This device is employed to assess and report on the presence of abnormal ECG states.
Change from baseline in the control rate of blood pressure (SBP/DBP <120/80 mm Hg) | baseline, six months
  The blood pressure was measured by a self-monitored electronic sphygmomanometer (Model Maibobo, Shenzhen Yike Network Technology Co., Ltd., China). The proportion of participants achieving a systolic blood pressure (SBP) below 120 mm Hg and a diastolic blood pressure (DBP) below 80 mm Hg is calculated by dividing the number of participants who meet these criteria by the total number of participants at baseline and each routine health check-up.
Change from baseline in SBP | baseline, six months
  The SBP is measured by a self-monitored electronic sphygmomanometer (Model Maibobo, Shenzhen Yike Network Technology Co., Ltd., China).
Change from baseline in DBP | baseline, six months
  The DBP was measured by a self-monitored electronic sphygmomanometer (Model Maibobo, Shenzhen Yike Network Technology Co., Ltd., China).
Change from baseline in left ventricular hypertrophy | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of left ventricular hypertrophy.
Change from baseline in sinus arrhythmia | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of sinus arrhythmia.
Change from baseline in right bundle branch block | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of right bundle branch block.
Change from baseline in ventricular premature beats | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of ventricular premature beats.
Change from baseline in atrial premature beats | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of atrial premature beats.
Change from baseline in Q waves | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of Q waves.
Change from baseline in T-wave changes | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of T-wave changes.
Change from baseline in ST changes | baseline, six months
  The trained staff use a handheld electrocardiographic recorder, CarePatch (ECG-H01, Hangzhou Proton Technology Co., Ltd., China) to measure the participants' the change of ST changes.
Change from baseline in the heat wave and cold spell perception score | baseline, six months
  The heat wave and cold spell perception score is measured by the heat wave and cold spell perception questionnaire. This questionnaire captures participants' perceptions of heatwave-related health risks and their level of preparedness. Respondents rate their responses on a continuous scale from 0 to 100, with 0 representing "not at all" or "very low" and 100 representing "very much" or "very high," allowing them to express the degree of their perception and concern.
Change from baseline in the PHQ-9 score | baseline, six months
  The PHQ-9 score is measured by Patient Health Questionnaire-9. This questionnaire evaluates nine key symptoms of depression experienced over the past two weeks, including loss of interest or pleasure in activities, feeling down or hopeless, trouble sleeping, fatigue, poor appetite or overeating, feelings of worthlessness or failure, difficulty concentrating, physical agitation or slowing, and thoughts of self-harm or suicide. Each symptom is rated on a scale from 0 (not at all) to 3 (nearly every day), with total scores ranging from 0 to 27. Scores of 5, 10, 15, and 20 indicate mild, moderate, moderately severe, and severe depression, respectively.
Change from baseline in the MMSE score | baseline, six months
  The MMSE score is measured by the mini-mental state examination. This examination evaluates five main areas: orientation (to time and place), memory (short-term and long-term), attention and calculation (concentration and basic arithmetic), language (fluency and comprehension), and executive function (complex task performance). Each area is scored on a scale from 0 to 5, with a total score ranging from 0 to 30. Typically, a score above 24 indicates normal cognitive function, while a score below 24 may suggest cognitive impairment.
Change from baseline in the GAD-7 score | baseline, six months
  The GAD-7 score is measured by the generalized anxiety disorder scale. This scale evaluates seven key symptoms of anxiety: feeling nervous, anxious, or on edge; not being able to stop or control worrying; worrying too much about different things; trouble relaxing; being so restless that it is hard to sit still; becoming easily annoyed or irritable; and feeling afraid as if something awful might happen. Each symptom is rated on a scale from 0 (not at all) to 3 (nearly every day), resulting in a total score ranging from 0 to 21. A score of 5 or above indicates the presence of generalized anxiety disorder symptoms, with higher scores reflecting greater symptom severity.
Change from baseline in the PSSS score | baseline, six months
  The PSSS score is measured by the perceived social support scale. This scale evaluates three key sources of support: family, friends, and significant others. It consists of 12 items, with four items each related to family, friends, and significant others. Participants rate their agreement with each statement on a scale from 1 (very strongly disagree) to 7 (very strongly agree), resulting in a total score ranging from 12 to 84, where higher scores indicate higher perceived social support.
Change from baseline in time-activity patterns | baseline, six months
  The time-activity patterns is measured by the self-reported time-activity diaries questionnaire. This questionnaire captures duration spent in various settings (such as outdoor environments, workplaces, transportation, home, and other indoor areas) and at different intensity levels of physical activity were recorded.
Change from baseline in HPSMBRS score | baseline, six months
  The HPSMBRS score is measured by the hypertension patient self-management behavior rating scale. The HPSMBRS consists of 33 individual items across six dimensions: medication management, condition monitoring, dietary management, exercise management, work-rest management, and emotional management. Each item is rated on a 1 to 5 Likert scale, with 1 indicating "never" and 5 indicating "always." The total score ranges from 33 to 165, with higher scores indicating better self-management. To ensure comparability across dimensions, individual scores are converted to standardized scores using the formula: standardized score = (actual ctual score of each factor / total score of each factor)×100. Self-management levels are categorized as low (<60), moderate (60~80), and high (>80) based on standardized scores.
Change from baseline in HPMARS score | baseline, six months
  The HPMARS score is measured by the hypertension patient medication adherence rating scale. The HPMARS consists of 8 individual items that assess key components of medication adherence: forgetting to take medication, intentional non-adherence, reducing or stopping medication due to side effects without consulting a doctor, forgetting medication during travel, forgetting to take medication the previous day, reducing dosage after symptoms are controlled, inconvenience of daily medication with maintaining adherence, and the frequency of forgetting to take medication. Each item is scored as 1 or 0, with the total HPMARS score ranging from 0 to 8. A total score of 8 indicates high adherence, 6 to 7 indicates moderate adherence, and a score below 6 suggests low adherence.
Changes in liver function biomarkers (e.g., albumin (ALB), alanine aminotransferase (ALT), aspartate aminotransferase (AST), etc.) from baseline | baseline, six months
  This section evaluates changes in liver function biomarkers using appropriate omics technologies to explore their potential role in liver-related diseases.
Changes in cardiovascular biomarkers (e.g., creatine kinase-MB (CK-MB), creatine kinase (CK), etc.) from baseline | baseline, six months
  This section assesses changes in cardiovascular function biomarkers through suitable omics techniques, investigating their involvement in cardiovascular diseases.
Changes in inflammatory biomarkers (e.g., interleukin-6 (IL-6), interleukin-1β (IL-1β), etc.) from baseline | baseline, six months
  This section examines the alterations in inflammatory biomarkers using relevant omics approaches, aiming to uncover their potential role in inflammatory and immune responses.
Changes in metabolic biomarkers (e.g., lactate dehydrogenase (LDH), high-density lipoprotein (HDL), low-density lipoprotein cholesterol (LDL) , etc.) from baseline | baseline, six months
  This section examines the alterations in metabolic biomarkers using relevant omics approaches, aiming to uncover their potential implications in metabolic processes and health outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Tiantian Li, Study Director — National lnstitute of Environmental Health, Chinese Center for Disease Controland Prevention
Locations (1):
- National Institute of Environmental Health, Chinese Center for Disease Control and Prevention, Beijing, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT06045403/Prot_SAP_000.pdf